CLINICAL TRIAL: NCT07247032
Title: Prospective Real World Heart Failure Management for Patient With CIED Remotely Monitored
Brief Title: Heart Failure Management for Patient With CIED Remotely Monitored
Acronym: PROACT-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Implicity (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A01507-42
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure With Reduced Ejection Fraction (HFrEF); Heart Failure With Decompensation; CRT and/or ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard remote monitoring (Active Comparator): Standard remote monitoring of ICD or CRT-D and standard remote monitoring of heart failure
  Interventions: Device: HF RM standard of care
- Remote monitoring with SmartSignalHF (Experimental): Remote monitoring with the SmartSignalHF device
  Interventions: Device: SmartSignalHF

INTERVENTIONS:
Device: SmartSignalHF — SmartSignalHF; a solution aiming to predict episodes of cardiac decompensation in patients implanted with an ICD or CRT-D
  Arms: Remote monitoring with SmartSignalHF
Device: HF RM standard of care — HF RM standard of care defined in the country (France or Germany)
  Arms: Standard remote monitoring

SUMMARY:
This randomized, controlled, open-label, parallel, multicenter clinical study evaluates the efficacy of SmartSignalHF compared with heart failure (HF) remote monitoring (RM) standard of care in implanted patients with heart failure. The primary objective is to determine whether SmartSignalHF reduces all-cause mortality and HF hospitalizations at 12 months.

DETAILED DESCRIPTION:
SmartSignalHF is a novel digital health solution designed to support clinical decision-making by continuously analyzing Cardiac Implantable Electronic Devices (CIED) and patient data and providing actionable alerts to healthcare teams. By integrating this digital solution into the remote monitoring of HF patients, the study aims to enhance early detection of decompensation events and optimize therapeutic treatments.

Eligible patients implanted with an Implantable Cardioverter Defibrillator (ICD) or a Cardiac Resynchronization Therapy Defibrillator (CRT-D) and diagnosed with chronic heart failure will be randomized in a 1:1 ratio to either SmartSignalHF remote monitoring solution or standard HF remote monitoring solution.

The primary endpoint is a composite of all-cause mortality and HF hospitalizations within 12 months after randomization. Secondary endpoints include individual components of the primary endpoint, quality-of-life measures, and adherence to guideline-directed medical therapy (GDMT).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-85
* Patient diagnosed with a New York Heart Association (NYHA) class II or III
* Patients with left ventricular ejection fraction ≼ 40 %
* Patient implanted with an ICD or CRT-D (BiV and/or LBBA pacing) since at least 30 days and compatible with SignalHF (Biotronik, Boston Scientific and Medtronic)
* Non-activation of others HF multisensor algorithms
* Patient remote monitored on Implicity CIED platform
* Patient with a documented diagnosis of heart failure, eligible to reimbursement in France or Germany for HF remote monitoring
* Patient is willing to be remotely monitored for heart failure
* HF treated according to European Society of Cardiology (ESC) guidelines

Exclusion Criteria:

* Patients undergoing or awaiting heart transplant or left ventricular assist device (LVAD) procedures
* Patients with a life expectancy of less than 12 months
* Patients enrolled in concurrent clinical studies
* Patients with a history of non-compliance with medical care or inability to comply with the study protocol
* Patients already receiving remote monitoring for heart failure
* Pregnant or breastfeeding women
* Subjects under legal protection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1132 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Composite measure of all-cause mortality and HF hospitalizations | From enrollment to the end of follow-up at 12 months

SECONDARY OUTCOMES:
All-cause mortality | From enrollment to the end of follow-up at 12 months
HF mortality | From enrollment to the end of follow-up at 12 months
HF hospitalizations | From enrollment to the end of follow-up at 12 months
HF readmissions | From enrollment to the end of follow-up at 12 months
HF outpatient visits | From enrollment to the end of follow-up at 12 months
All cause hospitalizations | From enrollment to the end of follow-up at 12 months
HF hospitalization duration | From enrollment to the end of follow-up at 12 months
Proportion of patients without contraindications receiving 4- drug GDMT | At 12 months
Proportion of patients achieving ≥ 50% target doses or maximum tolerated doses for each drug class | At 12 months
Proportion of patients achieving 100% target doses or maximum tolerated doses for each drug class | At 12 months
Minnesota Living with Heart Failure Questionnaire (MLHFQ) total score | At baseline and at 12 months
  The Minnesota Living With Heart Failure Questionnaire (MLHFQ) total score ranges from a minimum of 0 (best possible health-related quality of life) to a maximum of 105 (worst possible health-related quality of life).
Rate of patients who completed the study follow-up | At 12 months
Rate of premature study discontinuation due to withdrawal of consent for remote monitoring | From enrollment to the end of follow-up at 12 months
Data completion rate | At 12 months
Adverse events linked to the device during the follow-up | From enrollment to the end of follow-up at 12 months